CLINICAL TRIAL: NCT02764229
Title: A Multicenter Open-label Extension Study to Assess the Safety and Tolerability of LYC-30937-EC in Subjects With Active Ulcerative Colitis
Brief Title: Open-label Extension Study to Assess Safety and Tolerability of LYC-30937-EC in Subjects With Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy of test drug
Sponsor: Lycera Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYC-30937-2002; 2016-003633-26 (EudraCT Number)
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LYC-30937-EC (Experimental): LYC-30937-EC 25 mg by mouth once daily
  Interventions: Drug: LYC-30937-EC

INTERVENTIONS:
Drug: LYC-30937-EC — LYC-30937-EC 25 mg by mouth once daily

SUMMARY:
The purpose of this study is to allow subjects completing study LYC-30937-2001 the opportunity to receive LYC-30937-EC 25 mg.

DETAILED DESCRIPTION:
Subjects who complete the 8 week treatment period of the double-blind, placebo-controlled study LYC-30937-2001 will have the option of receiving LYC-30397-EC 25 mg PO QD in this open-label extension study (LYC-30937-2002). Subjects meeting eligibility criteria will enter this open-label extension trial upon completion of the LYC-30937-2001 Week 8 study procedures. This open-label extension study will consist of 44 weeks of treatment followed by a 2 weeks post-treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 8-week double-blind treatment period of study LYC-30937-2001
* Male and females of childbearing potential must agree to use adequate birth control during the study and for 30 days after discontinuing study drug
* Non-pregnant, non-lactating females who are not planning to become pregnant while enrolled in this study
* Investigator considers it safe and potentially beneficial to participate
* Ability to provide written informed consent and to be compliant with study schedule

Exclusion Criteria:

* Subjects who completed study LYC-30937-2001, but who experienced a serious adverse event that was considered related to investigational product, has an unstable medical condition, or for any other reason in the opinion of the investigator should not participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Jeffrey Wilkins, MD, Study Director — Lycera Corp.
Locations (33):
- United States (9):
  - Lycera Investigational Site, Little Rock, Arkansas
  - Lycera Investigational Site, Mission Hills, California
  - Lycera Investigational Site, Miami, Florida
  - Lycera Investigational Site, Chicago, Illinois
  - Lycera Investigational Site, Ann Arbor, Michigan
  - Lycera investigational site, Greenville, North Carolina
  - Lycera Investigational Site, Nashville, Tennessee
  - Lycera Investigational Site, Houston, Texas
  - Lycera investigational site, San Antonio, Texas
- Czechia (3):
  - Lycera Investigational Site, Ostrava
  - Lycera Investigational Site, Prague
  - Lycera Investigational Site, Ústí nad Labem
- Lycera Investigational Site, Budapest, Hungary
- Lycera Investigational Site, Rotterdam, Netherlands
- Poland (14):
  - Lycera Investigational Site, Bydgoszcz
  - Lycera Investigational Site, Katowice
  - Lycera Investigational Site, Kielce
  - Lycera Investigational Site, Krakow
  - Lycera Investigational Site, Lublin
  - Lycera Investigational Site, Piaseczno
  - Lycera Investigational Site, Poznan
  - Lycera Investigational Site, Skierniewice
  - Lycera Investigational Site, Sopot
  - Lycera Investigational Site, Staszów
  - Lycera Investigational Site, Szczecin
  - Lycera Investigational Site, Warsaw
  - Lycera Investigational Site, Wroclaw
  - Lycera Investigational Site, Włocławek
- Serbia (5):
  - Lycera Investigational Site, Belgrade
  - Lycera Investigational Site, Kragujevac
  - Lycera Investigational Site, Niš
  - Lycera Investigational Site, Subotica
  - Lycera Investigational Site, Zrenjanin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 40 study centers with the United States, Poland, Hungary, Czech Republic, Serbia and Netherlands. Study centers included academic medical centers and non-academic medical clinics.
Pre-assignment Details: Eligible subjects were those completing the preceding double-blind study LYC-30937-2001 Week 8 visit.
Period: Overall Study
Arm/Group | LYC-30937-EC
Started | 112
Completed | 10
Not Completed | 102
Not completed — Withdrawal by Subject | 15
Not completed — Adverse Event | 9
Not completed — Physician Decision | 5
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 1
Not completed — Study Stopped by Sponsor | 69

BASELINE CHARACTERISTICS:
Arm/Group | LYC-30937-EC
Number analyzed (Participants) | 112
Age, Continuous [Mean (Full Range); unit: years] | 41.5 [19 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 109
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: subjects] — Enrolled subjects were from Netherlands, Hungary, United States, Czechia, Poland, Serbia.
  subjects
    Netherlands | 3
    Hungary | 2
    United States | 22
    Czechia | 4
    Poland | 76
    Serbia | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Types of Adverse Events (AEs), Serious Adverse Events and AEs That Led to Discontinuation of Treatment
Description: Adverse events (AEs) were collected from the time a subject signed the informed consent and completed participation in the preceding double-blind trial LYC-30937-2001. Treatment-emergent adverse events (TEAEs) are AEs occurring or worsening after the first dose of study drug (LYC-30937-EC 25 mg). Adverse event severity was assessed by the Investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 4.03, with grading as follows: Grade 1 = mild (asymptomatic or mild symptoms), Grade 2 = moderate (minimal, local intervention, or noninvasive intervention indicated); Grade 3 = severe (or medically significant but not life-threatening); Grade 4 = life-threatening; Grade 5 = death.
Time Frame: 46 weeks
Population: Safety Set, consisting of all subjects who took at least 1 dose of study drug. 112 subjects signed consent to participate in the study and 111 of these were confirmed to have taken at least 1 dose of study drug. (One subject was lost to follow-up after enrolling and it was not confirmed that they took study drug.)
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC
Number analyzed (Participants) | 111
Participants
  Subjects with ≥ 1 AE | 56
  Subjects with ≥ 1 SAE | 6
  Subjects with AE leading to discontinuation | 9

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent through their last study visit, up to 46 weeks.
Description: Adverse events occurring after the first dose of study drug (treatment-emergent adverse events) are reported in this section.
Arm/Group | LYC-30937-EC
All-Cause Mortality (participants affected / at risk) | 0/111
Serious Adverse Events (participants affected / at risk) | 6/111
Other Adverse Events (participants affected / at risk) | 18/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYC-30937-EC (N=111)
Ulcerative colitis (Gastrointestinal disorders) | 2 (2) — exacerbation of existing ulcerative colitis
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Chronic obstructuve pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — exacerbation of existing COPD
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYC-30937-EC (N=111)
Colitis ulcerative (Gastrointestinal disorders) | 11 (15) — exacerbation of existing ulcerative colitis
Anaemia (Blood and lymphatic system disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center results cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then Investigator can publish if manuscript is submitted to Lycera ≥ 60 days prior to submission (or per Investigator contract). If Lycera decides publication would hinder development, Investigator must delay submission. Investigator must delete confidential information before submission and defer publication to allow patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT02764229/Prot_SAP_000.pdf